CLINICAL TRIAL: NCT00003599
Title: A Randomized Study of the Effect of Alpha-tocopherol (AT) on 13-cis-retinoic Acid (13-cRA) Toxicity in a Preliminary Chemoprevention Trial in Former and Current Smokers
Brief Title: Vitamin E in Preventing the Side Effects of Isotretinoin in Former and Current Smokers Who Are Receiving Isotretinoin to Prevent Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DM97-078; P30CA016672 (NIH); MDA-DM-97078 (Other: UT MD Anderson Cancer Center); NCI-P98-0132; CDR0000066672 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Vitamin E; alpha-Tocopherol; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Alpha-tocopherol (AT) orally and isotretinoin orally daily (arm I)
  Interventions: Dietary Supplement: Vitamin E (AT); Drug: Isotretinoin
- Arm II (Experimental): Isotretinoin orally plus AT placebo orally daily (arm II).
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Dietary Supplement: Vitamin E (AT) — Orally daily
  Other Names: alpha-tocopherol; AT
  Arms: Arm I
Drug: Isotretinoin — Orally daily
  Other Names: Accutane; 13-cis-Retinoic acid

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of isotretinoin may be an effective way to prevent lung cancer. Vitamin E may prevent the side effects of isotretinoin therapy.

PURPOSE: Randomized clinical trial to study the effectiveness of vitamin E in preventing the side effects of isotretinoin in former and current smokers who are receiving isotretinoin to prevent lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the addition of alpha-tocopherol (AT; vitamin E) to isotretinoin decreases the incidence of Grade II and higher toxicity of isotretinoin when administered to former and current smokers. II. Determine the compliance rate of isotretinoin of smoker and former smokers with or without AT over a six month period. III. Determine the feasibility of recruiting former and current smokers with or without AT over a six month period. IV. Determine the effect of isotretinoin administration on serum retinol and retinol-binding protein levels in these patients.

OUTLINE: This is randomized, placebo controlled study. Patients are stratified by smoking status (current smoker vs former smoker) and age (less than 50 vs 50 and over). Patients are randomized to be take alpha-tocopherol (AT) orally and isotretinoin orally daily (arm I) or isotretinoin orally plus AT placebo orally daily (arm II). Treatment in each arm continues for 6 months. Patients are followed at 1, 3, 6, and 7 months from start of treatment.

PROJECTED ACCRUAL: There will be 300 patients (150 per arm) accrued into this study over an estimated 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Current smokers with 20+ packs per year history of smoking OR Former smokers who discontinued smoking 1 year prior to registration (less than 5 cigarettes in the prior year) and had a 20+ packs per year history prior to discontinuing smoking

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 40 IU/mL OR SGPT less than IU/mL Renal: Not specified Other: Fasting triglycerides less than 320 mg/dL No prior malignancy in the past 5 years except nonmelanoma skin cancer or noninvasive cervical cancer No history of malabsorption syndrome Not pregnant Effective contraception required of all fertile persons

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior isotretinoin Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No prior warfarin or its derivatives At least 3 months since megadose vitamin A (greater than 25,000 IU/day) or beta-carotene greater than 30 mg/day or alpha-tocopherol at least 400 IU daily No concurrent megadose vitamin A (greater than 25,000 IU/day), beta-carotene greater than 30 mg/day, alpha-tocopherol at least 400 IU daily, or other daily supplements and tonics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Effect of Alpha-tocopherol (AT) on 13-cis-retinoic Acid (13-cRA) Toxicity | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rodger J. Winn, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org